CLINICAL TRIAL: NCT00344656
Title: The Study of Appetite-Related Brain Activity With Functional Magnetic Resonance Imaging in Women With Anorexia Nervosa
Brief Title: Appetite-Related Brain Activity in Women With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Other Study IDs: #4850
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Eating Disorders; Anorexia Nervosa
Keywords: Eating Disorders; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects and Controls: Patients with DSM-IV Anorexia Nervosa

SUMMARY:
This study will use functional magnetic resonance imaging to compare appetite-related brain activity in women with anorexia nervosa before and after receiving treatment for the disorder.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious eating disorder that is characterized by an extreme loss of appetite. People with AN view themselves as overweight and cannot bring themselves to eat, even though most are dangerously thin. Functional magnetic resonance imaging (fMRI) is a technique that can be used to determine which parts of the brain are activated by physical stimuli. When a certain stimulus is introduced, blood flow to the corresponding area of the brain increases. This increase in blood flow is depicted on the fMRI scan. A person with AN may have different responses to food when evaluated prior to treatment versus after treatment. This study will use fMRI to compare appetite-related brain activity in women with AN before and after receiving treatment for the disorder.

Participants in this study will undergo two fMRI scans. Participants with AN will have one scan before entering the "weight gain phase" of treatment for AN and another scan upon completion of treatment. Healthy volunteers will undergo scans during a similar time frame. Participants will not be allowed to eat from midnight on the night before the scan until after the fMRI procedure, but they may drink water. During the scan, participants will be shown various objects and real foods; they will also be asked to touch the objects and food with their eyes closed. Each visit will last approximately 45 minutes. Ear protectors will be provided to reduce scanner noise.

ELIGIBILITY:
Inclusion Criteria:

For Participants with AN:

* DSM-IV diagnosis of AN (restricting or binge eating/purging subtype)
* Medically stable (not continuing to lose weight and vital signs stable)

For Healthy Participants:

* Currently weighs 80-120% of ideal weight
* no history of binge eating disorder or vomiting
* no current or past psychiatric illness

Exclusion Criteria:

For Participants with AN:

* Currently taking medication
* Current substance abuse or dependence disorder
* History of suicide attempt or other self-injurious behavior within 6 months prior to study entry
* Non-removable metal on or inside the body (e.g., metal pacemaker, surgical clips, metallic-ink tattoos)

For Healthy Participants:

* Current or past psychiatric illness
* History of binge eating or vomiting
* Any significant medical or neurologic illness
* Currently taking medication
* History of drug or alcohol abuse within 3 months prior to study entry
* Non-removable metal on or inside the body (e.g., metal pacemaker, surgical clips, metallic-ink tattoos)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with AN between 18 and 45 years of age hospitalized for treatment of anorexia nervosa.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2004-10; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Mayer, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States